CLINICAL TRIAL: NCT06271928
Title: The Efficacy and Safety of Chinese Herbal Compound Yijing Keli in the Treatment of Ovarian Aging: A Multicenter and Prospective Study.
Brief Title: A Multicenter Clinical Study of Yijing Keli in the Treatment of Ovarian Aging
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jinjin Zhang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220634-yijingkeli
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Once enrolled, participants will be administrated Yijing Keli and followed by a 3-month medication cycle. The usage of this herbal compound is to take orally twice a day(two sacks per). Add it to about 200ml warm water and take it half an hour before breakfast in the morning and half an hour before bedtime in the evening except menstrual period.
  Interventions: Drug: Yijing Keli

INTERVENTIONS:
Drug: Yijing Keli — Once enrolled, participants will be administrated Yijing Keli

SUMMARY:
Ovarian aging (OA) seriously affects the physical and mental health of women. Nowadays, Chinese herbs have huge appeal and potential in treating OA. We have created a new Chinese herbal combination Yijing Keli, whereas its safety and efficacy still need to be validated. Hence, we will perform a population-based, multicenter study to confirm the safety and efficacy of Yijing Keli in therapy of OA. We aim to provide a solid evidence for TCM in therapy of OA.

ELIGIBILITY:
Inclusion Criteria:

1. The age range of patient is 18-55 years old.
2. The diagnostic criteria for ovarian aging.
3. Sign the informed consent form.

Exclusion Criteria:

1. Patient is known to be allergic or unsuitable for the Chinese herbal compound.
2. Women who are pregnant and lactating.
3. Abnormal uterine bleeding, except ovulation disorders.
4. Women is taking hormone drugs and has stopped taking them within 3 months;
5. Women with endometriosis, myadenosis, submucosal fibroids or the size of non- submucosal fibroids is more than 4 cm.
6. The nature of pelvic mass is unknown.
7. Women with polycystic ovary syndrome, hyperprolactinemia, hyperandrogenemia, diabetes, thyroid and adrenal dysfunction and other endocrine diseases affecting ovulation.
8. Patients with serious primary diseases such as cardiovascular, liver, kidney, lung, biliary, hematopoietic system (Hb<90g/L) and malignant tumor, and psychiatric patients.
9. Patients are participating in other clinical trials or have participated in other clinical trials within the last month.
10. Unsuitable for the study evaluated by the investigator.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
the recovery rate of ovarian function | 6 months
  evaluations of ovarian funtion are mainly based on the levels of AMH, basal serum FSH, and AFC. If the serum FSH level is lower than 10 mIU/mL, the serum AMH level is greater than 1.1 ng/mL, or AFC is more than 6 after treatment, it is considered effective. In addition, an improvement of more than 50% in these indicators after treatment can also be considered effective.

CONTACTS AND LOCATIONS:
Overall Officials: jinjin zhang, professor, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes